CLINICAL TRIAL: NCT04567238
Title: Impact of Reduced Cannabis Use on Functional Outcomes (R33 Phase)
Acronym: FOCUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00100100_1
Record Dates: First submitted 2020-09-23; First posted 2020-09-28 (Actual); Results first posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-11

CONDITIONS: Cannabis; Cannabis Use
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduced Use Condition (Experimental): Participants in the reduced use condition will be provided mobile contingency management, in which they are paid to provide marijuana saliva readings that suggest they have been abstinent from marijuana use.
  Interventions: Behavioral: Mobile contingency management
- Control Condition (No Intervention): Participants in the control condition will be asked to provide marijuana saliva readings, but they are not paid for abstinent readings. Instead, their payments are yoked to the average amount of payment made by two participants in the reduced use condition.

INTERVENTIONS:
Behavioral: Mobile contingency management — Mobile contingency management is a mobile-phone based behavioral therapy that provides positive reinforcement (i.e., money) for abstinence that is highly effective at reducing substance use.
  Other Names: mCM
  Arms: Reduced Use Condition

SUMMARY:
Nearly 20 million Americans report use of cannabis in the past month, and heavy cannabis use has increased by nearly 60% in the U.S. since 2007. Heavy cannabis use is associated with lower educational attainment, reduced physical activity, increased rates of addiction and unemployment, and neuropsychological deficits. Studies suggest that cannabis use is also associated with increased mental health symptoms, drugged driving, and traffic accidents. While there is evidence that sustained abstinence can lead to improvements in the functional outcomes of former users, the degree to which reductions alone (i.e., not sustained abstinence) in cannabis use might be associated with positive changes in functional outcomes is unknown. This is a critical gap in the literature, as many interventions for cannabis and other drugs are associated with decreases in frequency and quantity of use, but fail to achieve an effect on overall abstinence rates. The objective of the present research is to use ecological momentary assessment (EMA), a real-time, naturalistic data collection method, to prospectively study the impact of reduced cannabis use on functional outcomes in heavy cannabis users. Contingency management (CM) will be used to promote reductions in frequency and quantity of cannabis use. CM is an intensive behavioral therapy that is highly effective at producing short-term reductions in illicit drug use. We have recently developed a novel approach that leverages mobile technology and recent developments in cannabis testing. We have pilot-tested this approach with heavy cannabis users and found that it is an acceptable and feasible method. The present research will use this technology in conjunction with EMA methods to study the impact of reduced cannabis use on key functional outcomes. Our central hypothesis is that reductions in frequency and quantity of cannabis use will lead to positive changes in cannabis users' mental health, self-efficacy, physical activity, working memory, health-related quality of life, and driving behavior. The rationale for this research is that it will provide the first and only real-time data concerning the potential impact of reductions in cannabis use on functional outcomes. As such, the findings from the present research will directly inform ongoing efforts to include reductions in illicit drug use as a valid, clinically-meaningful outcome measure in clinical trials of pharmacotherapies for the treatment of substance use disorders.

ELIGIBILITY:
Inclusion Criteria:

* Report 40 or more days of cannabis use (other than ingested cannabis, i.e., edibles) in past 90 days
* Can speak and write fluent conversational English
* Are between 18 and 80 years of age
* Are willing to attempt to reduce frequency of cannabis use
* Complete at least 10 of the 14 nightly diaries during the ad lib phase of the study procedures.

Exclusion Criteria:

* Are expected to have an unstable medication regimen during the study
* Are currently receiving non-study treatment for cannabis use disorder
* Are pregnant or become pregnant
* Meet criteria for a serious mental illness (e.g., bipolar disorder, schizophrenia)
* Meet criteria for a substance use disorder other than nicotine or cannabis use disorders
* Are currently imprisoned or in psychiatric hospitalization or become imprisoned or in psychiatric hospitalization
* Report imminent risk for suicide or homicide
* Meet criteria for bio-verified sustained abstinence (i.e., all of their saliva tests are negative during the 6-week experimental phase of the study)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-11-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 76 participants were deemed eligible for the study at screen. Six participants were withdrawn, dropped out, or lost to contact during the ad lib phase of the study, so were not randomized to a study group. Ten participants didn't meet the 10 of 14 nightly diary minimum during the ad lib phase of the study, so were withdrawn prior to randomization.
Period: Overall Study
Arm/Group | Reduced Use Condition | Control Condition
Started | 40 | 20
Completed | 40 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: One participant was excluded from the analyses because the participant's reported mean daily cannabis use in grams was higher than five standard deviations of the rest of the sample, suggesting inaccurate reporting.
Groups:
- Total: Total of all reporting groups
Arm/Group | Reduced Use Condition | Control Condition | Total
Number analyzed (Participants) | 40 | 19 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (13.16) | 35.89 (14.34) | 38.1 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 15 | 40
  Male | 15 | 4 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 40 | 18 | 58
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 8 | 20
  White | 24 | 8 | 32
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 19 | 59

OUTCOME MEASURES:

1. Primary Outcome: Change in Mental Health Symptoms
Description: Mental health symptoms will be measured by the 90-item Symptom Checklist (SCL-90). This measure has a scoring range of 0 to 360, with lower scores indicating lower distress related to mental health.
Time Frame: Baseline and post-treatment (approximately eight weeks)
Population: Some participants were withdrawn from analyses due to missing data at the post-treatment visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reduced Use Condition | Control Condition
Number analyzed (Participants) | 38 | 15
score on a scale | -0.02 (0.31) | 0.11 (0.41)

2. Primary Outcome: Change in Self-reported Self-efficacy
Description: Self-efficacy will be measured by the Marijuana Reduction Strategies Self-Efficacy Scale. This measure has a scoring range of 0 to 84, with higher scores indicating increased self-efficacy.
Time Frame: Baseline and post-treatment (approximately eight weeks)
Population: Some participants were withdrawn from analyses due to missing data at the post-treatment visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reduced Use Condition | Control Condition
Number analyzed (Participants) | 34 | 15
score on a scale | -4.13 (56.40) | -16.07 (30.47)

3. Primary Outcome: Change in Physical Activity as Measured by the Leisure-Time Physical Activity Questionnaire
Description: Physical activity will be measured using the Leisure-Time Physical Activity Questionnaire. Scores range from 0 to 99, with higher scores indicating increased physical activity.
Time Frame: Baseline and post-treatment (approximately eight weeks)
Population: Some participants were withdrawn from analyses due to missing data at the post-treatment visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reduced Use Condition | Control Condition
Number analyzed (Participants) | 35 | 15
score on a scale | -0.46 (23.06) | 4.07 (16.05)

4. Primary Outcome: Change in Physical Activity as Measured by the International Physical Activity Questionnaire
Description: Physical activity will be measured using a continuous score on the International Physical Activity Questionnaire. The score is calculated by multiplying metabolic equivalents times minutes per day times days per week; scores range from 0 to 13,440. Higher scores indicate increased physical activity.
Time Frame: Time Frame: Baseline and post-treatment (approximately eight weeks)
Population: Some participants were withdrawn from analyses due to missing data at the post-treatment visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Reduced Use Condition | Control Condition
Number analyzed (Participants) | 34 | 11
units on a scale | -855.22 (5946.72) | -439.23 (5330.92)

5. Secondary Outcome: Change in Health-related Quality of Life, WHOQOL-BREF
Description: Health-related quality of life will be measured with the World Health Organization Quality of Life Brief (WHOQOL-BREF). The measure has a scoring range of 0 to 100, with higher scores indicating a higher quality of life.
Time Frame: Baseline and post-treatment (approximately eight weeks)
Population: Some participants were withdrawn from analyses due to missing data at the post-treatment visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reduced Use Condition | Control Condition
Number analyzed (Participants) | 37 | 14
score on a scale | 4.76 (14.77) | -1.93 (12.31)

6. Secondary Outcome: Change in Visual Working Memory
Description: Visual working memory will be measured by the Visual Working Memory (VWM) Index of Wechsler Memory Scale, which is comprised of the Symbol Span and Spatial Addition subtests, whose scores are added together to create a VWM score. Although this scale has no minimum or maximum score, higher scores indicate better visual working memory.
Time Frame: Baseline and post-treatment (approximately eight weeks)
Population: Some participants were withdrawn from analyses due to missing data at the post-treatment visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reduced Use Condition | Control Condition
Number analyzed (Participants) | 37 | 13
score on a scale | 1.95 (2.65) | -0.15 (3.44)

7. Secondary Outcome: Change in Auditory Working Memory
Description: Auditory working memory will be measured by the Auditory Working Memory (AWM) Index of Wechsler Memory Scale, which is comprised of the Digit Span and Letter-Number Sequencing subtests, whose scores are added together to create a AWM score. Although this scale has no minimum or maximum score, higher scores indicate better auditory working memory.
Time Frame: Baseline and post-treatment (approximately eight weeks)
Population: Some participants were withdrawn from analyses due to missing data at the post-treatment visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reduced Use Condition | Control Condition
Number analyzed (Participants) | 38 | 14
score on a scale | 0.74 (3.17) | -0.43 (2.59)

8. Secondary Outcome: Change in Impulsivity as Measured by Delay Discounting (i.e., Iowa Gambling Task)
Description: Impulsivity will be measured with a delay discounting task called the Iowa Gambling Task. Scores range from -100 to 100. Higher scores indicate more advantageous choices (i.e., lower impulsivity).
Time Frame: Baseline and post-treatment (approximately eight weeks)
Population: Some participants were withdrawn from analyses due to missing data at the post-treatment visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reduced Use Condition | Control Condition
Number analyzed (Participants) | 38 | 14
score on a scale | -5.89 (51.92) | -0.14 (30.92)

9. Secondary Outcome: Change in Impulsivity as Measured by the Balloon Analogue Risk Task
Description: Impulsivity will be measured with the Balloon Analogue Risk Task. Scores range from 0 to 128, and higher scores indicate higher impulsivity.
Time Frame: Baseline and post-treatment (approximately eight weeks)
Population: Some participants were withdrawn from analyses due to missing data at the post-treatment visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reduced Use Condition | Control Condition
Number analyzed (Participants) | 33 | 12
score on a scale | 5.58 (10.96) | 4.73 (6.09)

10. Secondary Outcome: Change in Impulsivity as Measured by Self-report
Description: Self-reported impulsivity will be measured with the Urgency, Premeditation (lack of), Perserverance (lack of), Sensation Seeking, Positive Urgency, Impulsive Behavior Scale (UPPS-P). The measure has a score range of 59 to 236. Higher scores indicate higher impulsivity.
Time Frame: Baseline and post-treatment (approximately eight weeks)
Population: Some participants were withdrawn from analyses due to missing data at the post-treatment visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Reduced Use Condition | Control Condition
Number analyzed (Participants) | 35 | 15
units on a scale | 1.16 (14.16) | 1.48 (13.18)

11. Secondary Outcome: Change in Number of Days of Drugged Driving
Description: Number of days of drugged driving in the past month will be self-reported by participants using a Timeline Follow-Back Interview.
Time Frame: Baseline and post-treatment (approximately eight weeks)
Population: Some participants were withdrawn from analyses due to missing data at the post-treatment visit.
Measure: Mean (Standard Deviation); unit: days per month
Arm/Group | Reduced Use Condition | Control Condition
Number analyzed (Participants) | 36 | 19
days per month | -6.44 (10.57) | -2.58 (7.73)

ADVERSE EVENTS:
Time Frame: 9 weeks
Arm/Group | Reduced Use Condition | Control Condition
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/19
Other Adverse Events (participants affected / at risk) | 0/40 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-16): https://cdn.clinicaltrials.gov/large-docs/38/NCT04567238/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-11): https://cdn.clinicaltrials.gov/large-docs/38/NCT04567238/ICF_001.pdf